CLINICAL TRIAL: NCT04409223
Title: A Phase III, Open Label, Randomised，Controlled, Multi-centre Study to Assess the Efficacy and Safety of Famitinib Versus Sunitinib in the Treatment of Advanced Gastrointestinal Stromal Tumour Patients After Failure of Imatinib
Brief Title: Efficacy and Safety of Famitinib Versus Sunitinib in the Treatment of Advanced Gastrointestinal Stromal Tumour Patients After Failure of Imatinib
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: R&D strategy adjustment
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1020-Ⅲ-303
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — famitinib; Sunitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Famitinib (Experimental)
  Interventions: Drug: Famitinib capsules
- Sunitinib (Active Comparator)
  Interventions: Drug: Sunitinib Capsules

INTERVENTIONS:
Drug: Famitinib capsules — Oral KIT/PDGFRA kinase inhibitor
  Arms: Famitinib
Drug: Sunitinib Capsules — Oral receptor tyrosine kinase (RTK) inhibitor
  Other Names: Sutent
  Arms: Sunitinib

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of famitinib in the treatment of advanced gastrointestinal stromal tumour patients after failure of imatinib compared to sunitinib.

ELIGIBILITY:
Inclusion Criteria:

1. The patients were enrolled voluntarily and signed informed consent, with good compliance and follow-up
2. Age ≥18 years (on the date of signing informed consent), for both men and women
3. Histologically confirmed metastatic or untreatable gastrointestinal stromal tumors have at least one measurable lesion that meets the criteria of RECIST v1.1. Lesions that have undergone radiotherapy must be confirmed by imaging to show progression after radiotherapy
4. Previous treatment with imatinib and eventual treatment failure (disease progression or toxicity intolerance during treatment)
5. The subjects were able to provide 10 ml blood samples and fresh or archived tumor tissue, or to receive biopsy at baseline for biomarker analysis.

   Note: if there is no archived tumor tissue sample, those at high risk of receiving biopsy after assessment by the researcher, who can provide the previous c-kit /PDGFRA test report, may also be selected for inclusion.
6. Eastern Cooperative Oncology Group performance status of 1 or lower
7. Expected survival ≥12 weeks
8. Vital organs and body functions meet the following requirements (no blood products or cell agents are allowed to be used within 14 days before the first use):

   Neutrophil absolute count ≥1.5×109/L; Platelet ≥ 100×109/L; Hemoglobin ≥ 90 g/L; Bilirubin ≤ 1.5×ULN; ALT and AST ≤2.5×ULN serum creatinine≤1.5×ULN; Results of urinary protein <2+; If urinary protein is ≥2+, 24-hour quantitative determination of urinary protein should be conducted, and no more than 1g/24 hour is qualified. Serum calcium, potassium, magnesium and phosphorus are within the normal range or have been corrected to the normal range before randomization. International standardized ratio INR≤ 1.5 and activated partial thromboplastin time APTT≤1.5×ULN; QTc≤ 450 ms (male), 470 ms (female); Left ventricular ejection fraction LVEF≥50%.
9. Use of a medically approved contraceptive method (e.g., intrauterine contraceptive device, contraceptive pill or condom) during the study period and within 90 days after the end of the study period for female patients of non-surgical sterilization or childbearing age; The serum HCG of female patients of childbearing age without surgical sterilization must be negative within 72 hours before randomization, and must be non-lactating to be enrolled; For male patients whose partners are women of childbearing age, effective methods of contraception should be used during the study period and within 90 days after the end of the study period.

Exclusion Criteria:

1. Previously received molecular targeted therapy for gastrointestinal stromal tumor except imatinib
2. The toxicity of previous imatinib or other treatments has not recovered or reached NCI CTC AE 5.0≤ 1
3. For patients with clinical symptoms of ascites or pleural effusion, those requiring puncture drainage or those who had received thoracic or ascites drainage within 1 month before signing informed consent were excluded, those with only small amount of ascites or pleural effusion on imaging but no clinical symptoms are qualified.
4. A second primary malignancy occurred within the last 5 years, except for adequately treated basal cell carcinoma, cutaneous squamous cell carcinoma, or carcinoma in situ of the cervix
5. Gastrointestinal stromal tumor with central nervous system metastasis
6. Inability to swallow, chronic diarrhea, intestinal obstruction, or factors that affect drug use and absorption
7. Bleeding≥ grade 2 occurred in the first 4 weeks of randomization (NCI, CTC, AE 5.0)
8. Symptoms occurred within 12 months before randomization: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass grafting, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or an arteriovenous embolism event (e.g., deep venous embolism of lower extremities, pulmonary embolism) within 6 months
9. There are clinical symptoms or diseases of the heart that are not well controlled, such as (1) heart failure above NYHA grade 2 (2) unstable angina (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention
10. Have hypertension, and cannot be well controlled by antihypertensive medication (systolic blood pressure ≥ 140mmhg or diastolic blood pressure ≥ 90mmhg, if the blood pressure was abnormal during the screening period, 2 consistent measurements must be done with an interval of more than 24h after medical correction); Previous hypertensive crisis or hypertensive encephalopathy;
11. Drug uncontrollable thyroid dysfunction
12. Known acute or chronic active hepatitis, HBV virus titer > 500 IU, HCV RNA detection > ULN
13. History of immunodeficiency, including HIV positive, acquired or congenital immunodeficiency disorder, or a history of organ transplantation
14. Major surgery or radiotherapy within the first 4 weeks of randomization, or temporary palliative radiotherapy for pain relief within the first 1 week of randomization; Molecular-targeted therapy (including oral targeted drugs in other clinical trials) is less than 5 drug half-lives away form randomization date
15. Participated in clinical trials of other drugs in the first 4 weeks of randomization
16. Digestive tract perforation occurred 3 months before randomization
17. In the judgment of the investigator, a concomitant illness (severe diabetes, a clear history of neurological or mental disorders, e.g., epilepsy or dementia) that seriously endangers the patient's safety or prevents the patient from completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 30 months
  Progression-free survival (PFS) assessed by BIRC based on RECIST 1.1 criteria

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 30 months
  Progression-free survival (PFS) assessed by BIRC based on mRECIST criteria
Progression-free survival (PFS) | 30 months
  Progression-free survival (PFS) assessed by researchers based on RECIST 1.1 criteria
time to disease progression (TTP) | 30 months
  Based on the RECIST v1.1 criteria, BIRC and the researchers' evaluation of: time to disease progression (TTP)
Time to treatment failure (TTF) | 30 months
  Based on the RECIST v1.1 criteria, BIRC and the researchers' evaluation of: Time to treatment failure (TTF);
Objective response rate (ORR) | 30 months
  Based on the RECIST v1.1 criteria, BIRC and the researchers' evaluation of: Objective response rate (ORR)
Duration of Response (DOR) | 30 months
  Based on the RECIST v1.1 criteria, BIRC and the researchers' evaluation of: Duration of Response (DOR)
Disease control rates (DCR) | 30 months
  Based on the RECIST v1.1 criteria, BIRC and the researchers' evaluation of: Disease control rates (DCR)
overall survival (OS) | 30 months
  Based on the RECIST v1.1 criteria, BIRC and the researchers' evaluation of: overall survival (OS)
Adverse Events and Serious Adverse Events | 30 months
  Adverse Events and Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, MD, Principal Investigator — Beijing 302 Hospital
Locations (1):
- 307 Hospital of PLA, Beijing, China